CLINICAL TRIAL: NCT02697266
Title: Individual Coping Strategies After Night Calls: Effects on Performing Clinical and Cognitive Tasks
Brief Title: The Effects of Night Call on Intellectual Performance
Status: Completed | Type: Observational
Sponsor: Haleh Saadat (Other)
Responsible Party: Sponsor-Investigator, Haleh Saadat, Director of Complementary and Alternative Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00143
Record Dates: First submitted 2015-12-21; First posted 2016-03-03 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post-call anesthesiologists: Attending anesthesiologists, and Anesthesiology residents
  Interventions: Other: No intervention
- Regular-shift anesthesiologists: Attending anesthesiologists, and Anesthesiology residents
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study.

SUMMARY:
The purpose of the current proposal will be to examine the clinical performance of both physicians in training as well as experienced faculty in pre and post call situations. Groups will be matched for gender, age, experience and employment duration during regular hours versus immediate post call hour.

DETAILED DESCRIPTION:
This is a prospective study evaluating the reaction time among attending anesthesiologists, and anesthesiology residents who take night shift call and are suffering from sleep deprivation. Investigators plan to examine clinical performance by measuring reaction times using a 10 minute psychomotor vigilance test device on physicians in training as well as experienced physicians in pre and post call situations.

All subjects will be informed of the scope and purpose of the study.

1. Attending Anesthesiologists: Gender, age, years of experience, years of employment at the institution, hours of sleep and circadian rhythm will be taken into effect.
2. Residents/Fellows: Gender, age, years of experience, years of employment at the institution and circadian rhythm will be taken into effect.

All study subjects will be asked to fill a questionnaire regarding demographic data, coping strategy Index.

1. Baseline instruments; including demographics, and coping strategy indicator (CSI), will be administrated.
2. Reaction time, mood and simple cognitive test will be measured at approximately 7 am of a regular day, (when the subject is not on call).
3. Reaction time, mood and simple cognitive test will be measured at approximately 7 am of after a call night.

This proposal attempts to examine the impact of night shift on mood, cognitive and motor task performance in physicians as compared to regular hours.

ELIGIBILITY:
Inclusion Criteria:

* Staff Attending Anesthesiologist who takes night shift call
* Anesthesiology residents who take night shift call

Exclusion Criteria:

* Staff unwilling to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty-four attending anesthesiologists and anesthesiology residents
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Reaction time | Regular Day and Post-call shifts - Through study completion, an average of one year.
  We plan to measure reaction times via a 10-minute psychomotor vigilance test (PVT, Ambulatory Monitoring Inc., NY) device. The PVT-192 Psychomotor Vigilance Task Monitor is a hand-held, self-contained system used for repetitive reaction time measurements.
Visual Analog Scale | Regular Day and Post-call shifts - Through study completion, an average of one year.
  Subjective sleepiness and alertness (and other parameters) will be measured via the Visual Analog Scale (VAS). This Questionnaire consists of several 100 millimeter lines, each of which is labeled at one end with the words "not at all" and the other end with the word "extremely". Centered under each line are the test adjectives which are as follows: "alert, able to concentrate, " anxious", "energetic", "feel confident", "irritable", "Jittery/nervous", "sleepy", and "talkative". The participants indicate the point on the line, which corresponded to the way they feel along the continuum at the time the test is taken. The score for each item consists of a number of millimeters from the left side of the line to the location at which the participants placed their mark.
Profile of mood states | Regular Day and Post-call shifts - Through study completion, an average of one year.
  Subjective evaluations of mood will be made with the Profile of Mood States (POMS). The POMS is a 65-Item questionnaire which, when scored according to the specific templates, measures affect or mood on scales: 1) Tension-Anxiety, 2) Depression-dejection, 3) anger-hostility, 4) vigor-activity, 5) fatigue-inertia, and 6) confusion-bewilderment. Factor scores on each scale will be analyzed.

SECONDARY OUTCOMES:
Coping Strategy Indicator (CSI): | Regular-shift - Through study completion, an average of one year.
  This is the self-report measure of three fundamental modes of coping that has demonstrated considerable psychometric strength. The CSI first instructs responders to select a recent stressful event from their lives and briefly describe it. Then, responders read a list of 33 specific coping behaviors, indicating the extent to which each was used to deal with the problem. Responders are summed to form three scales: problem solving, seeking social support and avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Haleh Saadat, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States